CLINICAL TRIAL: NCT05008055
Title: A Modular Phase II, Open-Label, Multicentre Study to Assess the Efficacy and Safety of Capivasertib in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (CAPITAL)
Brief Title: Study of Capivasertib in Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Acronym: CAPITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D361FC00001; 2021-000870-27 (EudraCT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-08-17 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Keywords: Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Capivasertib monotherapy
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Capivasertib monotherapy (Experimental): Participants with R/R FL, R/R MZL, and R/R MCL will receive capivasertib orally until progression of disease (PD) or unacceptable toxicity.
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — Capivasertib will be taken orally twice a day (BD) 4 days on/ 3 days off.

SUMMARY:
This study is an open-label, multicenter Phase II study of capivasertib administered orally in participants with Relapsed or Refractory (R/R) B-cell Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
The study protocol follows a modular design. The study will investigate the safety and efficacy of capivasertib monotherapy in participants with R/R Follicular Lymphoma (FL), Marginal Zone Lymphoma (MZL), and Mantle Cell Lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age, at the time of signing the informed consent
* Eastern Cooperative Oncology Group performance status ≤ 2
* Life expectancy > 6 months
* Female participants must not be breast-feeding and must have a negative pregnancy test (serum) prior to start of dosing

Module 1 specific inclusion criteria:

Additional Inclusion Criteria for Cohort 1A (R/R FL):

1. Histologically confirmed diagnosis of FL Grade 1, 2, or 3a as assessed by investigator or local pathologist
2. Current need for systemic treatment based on the Investigator's opinion
3. Relapsed, progressed or refractory (defined as failure to achieve at least a partial response [PR]) after at least 2 prior systemic lines of therapy (including anti-CD20 monoclonal antibody [mAb] and an alkylating agent)
4. Bi-dimensionally measurable disease on cross sectional imaging by computed tomography (CT) or magnetic resonance imaging (MRI) with at least one nodal lesion > 1.5 cm in the long axis or at least one extranodal lesion > 1 cm in long axis.

Additional Inclusion Criteria for Cohort 1B (R/R MZL):

1. Histologically confirmed MZL including splenic, nodal, and extranodal subtypes as assessed by investigator or local pathologist
2. Current need for systemic treatment based on the Investigator's opinion
3. Relapsed, progressed or refractory (defined as failure to achieve at least a PR) after at least 2 prior systemic lines of therapy (including at least one anti-CD20mAb directed regimen either as monotherapy or as chemoimmunotherapy; Helicobacter pylori eradication and radiation therapy alone will not be considered a systemic treatment regimen)
4. Bi-dimensionally measurable disease on cross sectional imaging by CT or MRI with at least one nodal lesion > 1.5 cm in the long axis or at least one extranodal lesion > 1 cm in long axis

Additional Inclusion Criteria for Cohort 1C (R/R MCL):

1. Histologically confirmed MCL, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1, as assessed by investigator or local pathologist
2. Relapsed, progressed or refractory (defined as failure to achieve at least a PR) after at least 2 prior systemic lines of therapy
3. Participants must have received as prior therapies

   Prior regimens must have included:
   * BTK inhibitor and
   * Anti-CD20mAb therapy
4. Bi-dimensionally measurable disease on cross sectional imaging by CT or MRI with at least one nodal lesion > 1.5 cm in the long axis or at least one extranodal lesion > 1 cm in long axis

Exclusion Criteria:

* Prior malignancy (other than the disease under study), except for adequately treated basal cell or squamous cell skin cancer, in situ cancer, or other cancer from which the participant has been disease free for ≥ 2 years
* With the exception of alopecia, any unresolved non-haematological toxicities from prior therapy ≥ Common Terminology Criteria for Adverse Events Grade 2 at the time of starting study treatment
* Known medically apparent central nervous system lymphoma or leptomeningeal disease
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values at screening:

  1. Absolute neutrophil count < 1.0 × 10^9/L; < 0.75 × 10^9/L in participants with known bone marrow involvement of malignant disease
  2. Platelets < 75 × 10^9/L; < 50 × 10^9/L in participants with known bone marrow involvement of malignant disease
  3. Creatinine clearance < 50 mL/min per the Cockcroft and Gault formula
* Clinically significant abnormalities of glucose metabolism as participants with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment and Glycosylated haemoglobin ≥ 8.0% (63.9 mmol/mol)
* Prior treatment with any of the following:

  1. Any investigational agents or study drugs from a previous clinical study within 5 half lives or 2 weeks from the first dose of capivasertib in this study
  2. Strong inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort), or drugs that are sensitive to inhibition of CYP3A4 within 1 week prior to the first dose of study treatment
  3. Prior allogenic Haematopoietic stem cell transplant (HSCT) within 6 months from the first dose of capivasertib (patients > 6 months after allogenic HSCT are eligible in the absence of active graft-versus-host disease and concomitant immune suppressive therapy). Prior cellular therapies (eg, Chimeric antigen receptor T therapy) and/or autologous HSCT within 3 months from the first dose of capivasertib
  4. Receipt of live, attenuated vaccine within 28 days before the first dose of study treatment(s)
  5. Participants who, due to other medical conditions /prior history /concomitant medications are, in the investigator's opinion, at a risk of a venous thromboembolism (VTE) and are not willing to accept the VTE prophylaxis, will be excluded. The initiation of an adequate VTE prophylaxis will be based on treating physician risk/benefit assessment and in agreement with the local management guidelines

Additional exclusion core criteria may apply, please refer to the protocol

Module 1 specific exclusion criteria:

1. Follicular lymphoma grade 3B
2. Known transformation to aggressive lymphoma, eg, large cell lymphoma
3. Participants who, in the Investigator's opinion, require immediate cytoreductive therapy for disease control

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (3):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Houston, Texas
- Research Site, Victoria, British Columbia, Canada
- Research Site, Aarhus N, Denmark
- France (2):
  - Research Site, Poitiers
  - Research Site, Villejuif
- South Korea (2):
  - Research Site, Busan
  - Research Site, Seoul
- Spain (3):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D361FC00001&attachmentIdentifier=de0ae606-15d1-4c8f-800e-5e67fdc17ac0&fileName=Capital_SAP_redacted_22_Nov_2023_English_D361FC00001.pdf&versionIdentifier=
- See also: Redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D361FC00001&attachmentIdentifier=780d4972-0b22-49a5-a776-7d0d2b0d922a&fileName=CAPITAL_CSP_redacted_24_Feb_2022_English_D361FC00001.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D361FC00001&attachmentIdentifier=7391f9ec-950d-44af-9363-9444687ed7ed&fileName=AZ_D361FC00001_(PXL_256606)_CSR_Synopsis_08_Mar_2024_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 3 November 2021 and analyses presented in this results form are based on a data cut-off of 22 August 2023.
Pre-assignment Details: Patients who met the inclusion and none of the exclusion criteria were enrolled to the study. This study consisted of a screening period of 28 days. All the study assessments were performed as per schedule of assessment.
Groups:
- Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy: Patients with R/R FL received capivasertib 480 mg orally until progression of disease (PD) or unacceptable toxicity, or if the patient/investigator requests to stop the treatment.
- Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy: Patients with R/R MZL received capivasertib 480 mg orally until PD or unacceptable toxicity, or if the patient/investigator requests to stop the treatment.
- Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy: Patients with R/R MCL received capivasertib 480 mg orally until PD or unacceptable toxicity, or if the patient/investigator requests to stop the treatment.
Period: Overall Study
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Started | 16 | 4 | 10
Completed | 13 | 3 | 9
Not Completed | 3 | 1 | 1
Not completed — Patients ongoing treatment at data cut-off date of 22 August 2023. | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included for baseline characteristics, and it included all patients who received any amount of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy | Total
Number analyzed (Participants) | 16 | 4 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (12.07) | 66.8 (4.92) | 76.2 (9.72) | 64.0 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 4 | 13
  Male | 9 | 2 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 0 | 0 | 5
  White | 10 | 3 | 7 | 20
  Other | 0 | 1 | 1 | 2
  Not reported | 1 | 0 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 12 | 4 | 5 | 21
  Missing | 0 | 0 | 4 | 4
  Other | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is defined as the proportion of patients achieving either complete response (CR) or partial response (PR) according to the Lugano 2014 Classification for non-Hodgkin lymphoma (NHL) as assessed by blinded independent central review (BICR).
Time Frame: First dose until progression of disease [PD] or last evaluable assessment in the absence of progression or data cut-off date (21.6 Months)
Population: Response evaluable analysis set included all patients, treated with study treatment, with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 16 | 3 | 10
Percentage of Patients | 18.8 [4.0 to 45.6] | 33.3 [0.8 to 90.6] | 30.0 [6.7 to 65.2]

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of first documented response until date of documented progression according to the Lugano 2014 Classification for NHL as assessed by BICR, or death due to any cause.
Time Frame: First documented response until date of documented progression or data-cut off date (21.6 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 3 | 1 | 3
Months | 1.9 [1.7 to NA] — The values were not calculable due to low number of patients. | NA [NA to NA] — The values were not calculable due to low number of patients. | 1.9 [NA to NA] — The values were not calculable due to low number of patients.

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the date of first dose until documented disease progression according to the Lugano 2014 Classification for NHL as assessed by BICR, or death due to any cause. The analysis included all dosed patients, regardless of whether the patient withdrew from therapy, received another anti lymphoma therapy, or clinically progressed prior to progression according to the Lugano 2014 Classification for NHL.
Time Frame: First dose until documented disease progression or data cut-off date (21.6 Months)
Population: Safety analysis set included all patients who received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 16 | 4 | 10
Months | 5.4 [3.4 to NA] — The upper limit of the 95% confidence interval (CI) was not reached due to the insufficient number of patients with events, and the short duration of follow-up. | NA [1.4 to NA] — The upper limit of the 95% CI was not reached due to the insufficient number of patients with events, and the short duration of follow-up. | 1.9 [0.9 to NA] — The upper limit of the 95% CI was not reached due to the insufficient number of patients with events, and the short duration of follow-up.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from the date of first dose until the date of death due to any cause. The analysis included all dosed patients, regardless of whether the patient withdrew from therapy or received another anti lymphoma therapy. Patients who had not died by the analysis DCO date were censored at their last known date of being alive before the DCO date. Patients who were known to be alive or dead after the DCO date were censored at the DCO date. Patients who were lost to follow-up were censored at the date when they were last known to have been alive.
Time Frame: First dose until data cut-off date (21.6 Months)
Population: Safety analysis set included all patients who received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 16 | 4 | 10
Months | NA [NA to NA] — Median and 95% CI could not be calculated as no patients were seen to experience the event of interest due to short duration of follow-up. | NA [1.4 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached. | NA [2.0 to NA] — The median and upper limit of 95% CI could not be calculated as they were not reached.

5. Secondary Outcome: Number of Patients With Adverse Events and Serious Adverse Events
Description: The safety and tolerability of the capivasertib treatment in each Cohort was assessed.
Time Frame: Screening (Day -28 to -1) until Post-treatment follow-up up to 30 days after last dose or long-term follow-up or study completion (Every 12 weeks until death or lost to follow-up, unless patient have withdrawn consent [up to 21.6 Months])
Population: Safety analysis set included all patients who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 16 | 4 | 10
Participants
  Any adverse event (AE) | 16 | 3 | 10
  Any AE possibly related to treatment | 14 | 3 | 8
  Any AE of CTCAE grade 3 or higher | 7 | 1 | 7
  Any AE of CTCAE grade 3 or higher, possibly related to treatment | 3 | 1 | 5
  Any AE with outcome = death | 0 | 0 | 0
  Any AE with outcome = death, possibly related to treatment | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 2 | 0 | 3
  Any SAE (including events with outcome = death), possibly related to treatment | 0 | 0 | 3

6. Secondary Outcome: Plasma Concentration of Capivasertib Overtime
Description: The plasma concentration of capivasertib when administered in patients in each Cohort was determined.
Time Frame: Cycle 1 (28-day treatment Cycle) Day 1 and on Cycle 1 Day 8, Cycle 1 Day 15 and Cycle 1 Day 22 (Pre-dose and post-dose)
Population: Pharmacokinetic (PK) analysis set included all patients who received at least 1 dose of capivasertib, for whom there is at least 1 reportable PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
Number analyzed (Participants) | 16 | 4 | 9
ng/mL
  Cycle 1 Day 1 (Post-dose [1 hour]): number analyzed (Participants) | 16 | 3 | 9
  Cycle 1 Day 1 (Post-dose [1 hour]) | 394.9 (157.0) | 414.4 (125.7) | 287.1 (676.2)
  Cycle 1 Day 1 (Post-dose [2 hours]): number analyzed (Participants) | 15 | 4 | 8
  Cycle 1 Day 1 (Post-dose [2 hours]) | 883.7 (59.12) | 962.9 (40.33) | 976.1 (58.27)
  Cycle 1 Day 1 (Post-dose [4 hours]): number analyzed (Participants) | 16 | 4 | 8
  Cycle 1 Day 1 (Post-dose [4 hours]) | 528.5 (49.28) | 677.2 (65.77) | 780.1 (56.99)
  Cycle 1 Day 8 (Pre-dose): number analyzed (Participants) | 15 | 4 | 5
  Cycle 1 Day 8 (Pre-dose) | 6.149 (207.4) | 8.477 (103.9) | 14.31 (138.8)
  Cycle 1 Day 15 (Pre-dose): number analyzed (Participants) | 14 | 4 | 3
  Cycle 1 Day 15 (Pre-dose) | 5.844 (146.1) | 9.245 (73.63) | 32.36 (373.5)
  Cycle 1 Day 22 (Pre-dose): number analyzed (Participants) | 12 | 2 | 2
  Cycle 1 Day 22 (Pre-dose) | 7.974 (372.2) | NA (NA) — Geometric mean was not quantified because in given time point, when less than or equal to 50% of the concentration values were not measurable or quantified. | NA (NA) — Geometric mean was not quantified because in given time point, when less than or equal to 50% of the concentration values were not measurable or quantified.

ADVERSE EVENTS:
Time Frame: Screening (Day -28 to -1) until Post-treatment follow-up up to 30 days after last dose or long-term follow-up or study completion (Every 12 weeks until death or lost to follow-up, unless patient have withdrawn consent [up to 21.6 Months])
Arm/Group | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/4 | 2/10
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/4 | 3/10
Other Adverse Events (participants affected / at risk) | 16/16 | 3/4 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy (N=16) | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy (N=4) | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy (N=10)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed or Refractory Follicular Lymphoma (R/R FL): Capivasertib Monotherapy (N=16) | Relapsed or Refractory Marginal Zone Lymphoma (R/R MZL): Capivasertib Monotherapy (N=4) | Relapsed or Refractory Mantle Cell Lymphoma (R/R MCL): Capivasertib Monotherapy (N=10)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (29) | 2 (3) | 4 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (6)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (5) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT05008055/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT05008055/SAP_001.pdf